CLINICAL TRIAL: NCT02325830
Title: The REDUCE FMR Trial: Safety and Efficacy of the Carillon Mitral Contour System® in Reducing Functional Mitral Regurgitation (FMR) Associated With Heart Failure
Brief Title: Carillon Mitral Contour System® for Reducing Functional Mitral Regurgitation
Acronym: REDUCE FMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiac Dimensions Pty Ltd (Industry)
Collaborators: Menzies Institute for Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVP 1627-01
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Results first posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-02

CONDITIONS: Mitral Valve Insufficiency; Heart Failure
Keywords: Functional mitral regurgitation; Secondary mitral regurgitation; Percutaneous mitral repair
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure

STUDY DESIGN:
Intervention Model Description: With crossover for sham procedure patients who are eligible at time of 12 month follow up.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Implantation of the Carillon Mitral Contour System
  Interventions: Device: Carillon Mitral Contour System
- Control Group (No Intervention): Optimized stable medical therapy

INTERVENTIONS:
Device: Carillon Mitral Contour System — Percutaneous mitral valve repair
  Arms: Treatment Group

SUMMARY:
The objective of this prospective, multi-center, randomized, double-blind trial is to assess the safety and efficacy of the Carillon Mitral Contour System in treating functional mitral regurgitation (FMR) associated with heart failure, compared to a randomized Control group which is medically managed according to heart failure guidelines.

DETAILED DESCRIPTION:
The American Heart Association (AHA) estimates that there are more than 22 million people worldwide with heart failure. Functional mitral regurgitation, defined as the leakage of the mitral valve caused by global or regional changes in left ventricular geometry as well as mitral annular dilation, occurs as a consequence of heart failure. Cardiac Dimensions has developed proprietary technology designed to address functional mitral regurgitation in a minimally invasive manner.

Cardiac Dimensions plans to conduct a clinical trial of the Carillon Mitral Contour System in study subjects with functional mitral regurgitation. This study is a prospective, randomized parallel-group, double-blind, multi-center clinical trial designed to examine the safety and efficacy of the Carillon Mitral Contour System in study subjects with functional mitral regurgitation. The study will consent up to 180 subjects in order to randomize up to 120 subjects at 25 investigational sites in Europe and Australia/New Zealand. Subjects will be randomized into one of two study groups using a 3:1 (Treatment group : Control group) ratio.

Study subjects who are eligible for this clinical study and have consented to participating in the study will undergo multiple assessments prior to randomization to evaluate the eligibility (inclusion/exclusion) criteria. Subjects who meet all eligibility criteria will be randomized into one of two study groups (Treatment or Control).

Study subjects randomized to the Treatment group will undergo a venous angiogram to assess the suitability of the coronary sinus/great cardiac vein (CS/GCV) for placement of the Carillon implant. If the subject meets the anatomic requirements for device placement, the Carillon implant procedure begins. With the distal aspect of the device anchored, incremental tension will be applied to plicate the peri-annular tissue. A transesophageal or transthoracic echocardiogram will be obtained during the procedure to evaluate the effect on functional mitral regurgitation and to evaluate left ventricular function. After the proximal anchor of the implant is locked in place, safety (including assessment of coronary arterial flow) and efficacy will be reconfirmed prior to releasing the Carillon implant from the delivery system.

Subjects randomized to the Control group will experience an index procedure similar to the Treatment group, however, without device placement. To ensure that subjects randomized to the Control group will not be able to deduce the treatment assignment based on the type of intervention or time associated with the procedure, minimal interventional procedures, such as femoral arterial pressure monitoring and a jugular venous drip. If a recent (within the last 3 months for ischemic cardiomyopathy or 12 months for non-ischemic cardiomyopathy) coronary angiogram is available, this assessment may be precluded.

After the study subjects are discharged, the subjects' primary care specialists (cardiologist/heart failure physician) and clinical investigation site staff will coordinate follow-up evaluations. Subjects will be evaluated at one (1), six (6), and twelve (12) months post-implant, to assess long-term safety, and functional and clinical status. (Reference Section 3.8-Study Follow-up Evaluations)

This study will provide for an independent Clinical Events Committee (CEC) and an independent Data Safety Monitoring Board (DSMB). The CEC will be responsible for adjudicating complications reported during the study that are related to study endpoints (objectives), the procedure or the device. The DSMB will review the safety data against the established criteria and in the context of other safety data accumulated to date and the continued validity of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dilated ischemic or non-ischemic cardiomyopathy
* Functional Mitral Regurgitation: 2+ (Moderate), 3+ (Moderate/Severe), or 4+ (Severe)
* New York Heart Association (NYHA) II, III, or IV
* Six Minute Walk distance of at least 150 meters and no farther than 450 meters
* Left Ventricular Ejection Fraction ≤ 50 %
* LV end diastolic dimension (LVEDD) >55mm or LVEDD/Body Surface Area (BSA) > 3.0cm/m2
* Stable heart failure medication regimen for at least three (3) months prior to index procedure

Exclusion Criteria:

* Hospitalization in past three (3) months due to myocardial infarction, coronary artery bypass graft surgery, and/or unstable angina
* Hospitalization in the past 30 days for coronary angioplasty or stent placement
* Subjects expected to require any cardiac surgery within one (1) year
* Subjects expected to require any percutaneous coronary intervention within 30 days of enrollment
* Pre-existing device (e.g., pacing lead) in coronary sinus (CS) / great cardiac vein (GCV), or anticipated need for CRT within twelve (12) months
* Presence of a coronary artery stent under the CS / GCV in the implant target zone
* Presence of left atrial appendage (LAA) clot.
* Presence of primary renal dysfunction or significantly compromised renal function as reflected by a serum creatinine > 2.2 mg/dL OR eGFR < 30 ml/min
* Inability to undertake a six-minute walk test due to physical restrictions/limitations
* Chronic severe pathology limiting survival to less than 12-months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2015-08-22 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2020-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horst Sievert, MD, Principal Investigator — Cardio Vascular Center; David Kaye, MD, Principal Investigator — The Alfred
Locations (31):
- Australia (6):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Prince Alfred, Sydney, New South Wales
  - Flinders Medical Centre, Adelaide, South Australia
  - Monash Health, Clayton, Victoria
  - Alfred Health, Prahran, Victoria
  - Prince Charles, Brisbane
- Czechia (3):
  - Olomouc University Hospital, Olomouc
  - Institut klinické a experimentální medicíny (IKEM), Prague
  - Na Homolce Hospital, Prague
- France (7):
  - Pôle Sante République, Clermont-Ferrand, Auvergne
  - Hôpital Privé Saint-Martin, Caen
  - Clinique du Millénaire, Montpellier
  - European Hospital Georges Pompidou, Paris
  - Clinique Saint-Hilaire, Rouen
  - Hôpital Charles Nicolle, Rouen
  - CHU Rangueil, Toulouse
- Germany (9):
  - Märkische Kliniken GmbH, Klinikum Lüdenscheid, Lüdenscheid, North Rhine-Westphalia
  - Charité Universitätsmedizin Berlin, Berlin
  - Augusta Kranken-Anstalt GmbH, Bochum
  - Cardio Vascular Center Frankfurt, Frankfurt
  - Klinikum Frankfurt Höchst GmbH, Frankfurt
  - University Hospital Frankfurt, Frankfurt am Main
  - Universitäts-Herzzentrum Freiburg, Freiburg im Breisgau
  - Sana Kliniken Lübeck, Lübeck
  - Elisabeth Krankenhaus GmbH, Recklinghausen
- Maastricht University Medical Centre, Maastricht, Netherlands
- Auckland City Hospital, Grafton, New Zealand
- Poznan University of Medical Sciences, Poznan, Poland
- United Kingdom (3):
  - Harefield Hospital, Harefield, Middlesex
  - Leeds Teaching Hospitals NHS Trust, Leeds, Yorkshire
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schofer J, Siminiak T, Haude M, Herrman JP, Vainer J, Wu JC, Levy WC, Mauri L, Feldman T, Kwong RY, Kaye DM, Duffy SJ, Tubler T, Degen H, Brandt MC, Van Bibber R, Goldberg S, Reuter DG, Hoppe UC. Percutaneous mitral annuloplasty for functional mitral regurgitation: results of the CARILLON Mitral Annuloplasty Device European Union Study. Circulation. 2009 Jul 28;120(4):326-33. doi: 10.1161/CIRCULATIONAHA.109.849885. Epub 2009 Jul 13. PMID 19597051
- [Background] Siminiak T, Wu JC, Haude M, Hoppe UC, Sadowski J, Lipiecki J, Fajadet J, Shah AM, Feldman T, Kaye DM, Goldberg SL, Levy WC, Solomon SD, Reuter DG. Treatment of functional mitral regurgitation by percutaneous annuloplasty: results of the TITAN Trial. Eur J Heart Fail. 2012 Aug;14(8):931-8. doi: 10.1093/eurjhf/hfs076. Epub 2012 May 21. PMID 22613584
- [Background] Siminiak T, Hoppe UC, Schofer J, Haude M, Herrman JP, Vainer J, Firek L, Reuter DG, Goldberg SL, Van Bibber R. Effectiveness and safety of percutaneous coronary sinus-based mitral valve repair in patients with dilated cardiomyopathy (from the AMADEUS trial). Am J Cardiol. 2009 Aug 15;104(4):565-70. doi: 10.1016/j.amjcard.2009.04.021. Epub 2009 May 29. PMID 19660613
- [Derived] Witte KK, Lipiecki J, Siminiak T, Meredith IT, Malkin CJ, Goldberg SL, Stark MA, von Bardeleben RS, Cremer PC, Jaber WA, Celermajer DS, Kaye DM, Sievert H. The REDUCE FMR Trial: A Randomized Sham-Controlled Study of Percutaneous Mitral Annuloplasty in Functional Mitral Regurgitation. JACC Heart Fail. 2019 Nov;7(11):945-955. doi: 10.1016/j.jchf.2019.06.011. Epub 2019 Sep 11. PMID 31521683

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 163 subjects consented to randomize 120. 28 Screen Failed prior to procedure 15 Excluded at the procedure due to angiographic results
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 87 | 33
Completed | 70 | 24
Not Completed | 17 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 87 | 33 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (9.7) | 69.1 (8.9) | 69.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 9 | 33
  Male | 63 | 24 | 87
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
NYHA [Count of Participants; unit: Participants] — Patients underwent physical exam including NYHA assessment at 1M, 6M, and 12M. Protocol definitions used for the study were consistent with NYHA classifications:
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g., walking short distances (20-100 m). Comfortable only at rest. Worse than Class II.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients. Worse than Class III.
  Participants
    NYHA II Mild symptoms | 39 | 16 | 55
    NYHA III Marked limitation | 46 | 17 | 63
    NYHA IV Severe limitations | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline Regurgitant Volume Associated With the Carillon Device Relative to the Control Population at 12 Months
Description: The primary echocardiographic index and primary endpoint of the REDUCE FMR study was Regurgitant Volume (RV) in the ITT population (N=120). RV was analyzed for the ITT patient population calculated as the mean change per randomization group among subjects with evaluable data. Between group comparisons were performed using the Students' t-test.
Time Frame: Baseline and 12 months
Population: Image quality from sites reduced ultimate number of images able to be analyze by central review committee for RV values.
Measure: Mean (95% Confidence Interval); unit: ml/beat
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 55 | 13
ml/beat | -7.07 [-11.68 to -2.46] | 3.32 [-5.98 to 12.62]

2. Primary Outcome: Difference in the Rate of Major Adverse Events Between Treatment (Carillon) and Control Groups
Description: Cumulative number of events for Death, Myocardial Infarction, Cardiac Perforation, Device embolization, and surgical or percutaneous intervention related to device.
Time Frame: Baseline and 12 months
Population: 120 randomized subjects, regardless of follow-up period.
Measure: Mean (95% Confidence Interval); unit: Mitral Regurgitant Volume (mL)
Groups:
- Treatment Group: Implantation of the Carillon Mitral Contour System Carillon Mitral Contour System: Percutaneous mitral valve repair
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 87 | 33
Mitral Regurgitant Volume (mL) | -7.07 [-11.68 to -2.46] | 3.32 [-5.98 to 12.62]

3. Secondary Outcome: Rate of Heart Failure Hospitalizations Between Treatment (Carillon) and Control Groups
Description: A diagnosis of acute decompensated heart failure hospitalization (ADHF) requires an in-hospital stay that includes at least one calendar date change and requires intravenous or mechanical heart failure treatment. The length of hospital stay will be calculated from admission to discharge to home or other disposition.
  The diagnosis of ADHF will be based on:
  * Symptoms of worsening heart failure such as increased shortness of breath, orthopnea, paroxysmal nocturnal dyspnea, fatigue, decreased exercise tolerance or history of weight gain;
  * Physical examination evidence such as neck vein distention, the presence of a third heart sound, bilateral pulmonary rales, worsening ascites or pedal edema, hypotension or signs of worsening end-organ perfusion; and/or
  * Laboratory evidence, which may include pulmonary congestion on chest x-ray, elevated natriuretic peptide level, worsening oxygenation or respiratory acidosis.
Time Frame: Baseline and 12 months
Population: Randomized subjects, per treatment arm
Measure: Mean (95% Confidence Interval); unit: Rate of HFH per patient-year
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 87 | 33
Rate of HFH per patient-year | 0.57 [0.41 to 0.72] | 0.73 [0.44 to 1.03]

4. Secondary Outcome: Change in Six-minute Walk Distance Between Treatment (Carillon) and Control Groups
Description: Subjects had 6-MWT conducted at baseline and each follow-up visit. The subject walked as far as they could within a 6-minute period. They were allowed to rest. The distance (in whole meters) was captured at each visit.
Time Frame: Baseline and 12 Months
Population: Randomized subjects
Measure: Mean (95% Confidence Interval); unit: Meters
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 87 | 33
Meters | 32.0 [-10.0 to 70] | 17.5 [-20.0 to 46.5]

5. Secondary Outcome: Change in Left Ventricular Volumes Between Treatment (Carillon) and Control Groups
Description: The volume of the left ventricle will be measured by a blinded echosonographer ajdn submitted to the core lab for blinded analysis. The ventricle will be measured as systole and diastole.
Time Frame: Baseline and 12 Months
Population: Randomized population with paired images from baseline to 12-month only.
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 47 | 16
mL
  LVEDV | -10.42 [-18.18 to -2.37] | 6.54 [-5.14 to 18.22]
  LVESV | -6.19 [-12.78 to 0.39] | 6.1 [-1.42 to 13.63]

ADVERSE EVENTS:
Time Frame: Adverse Event Data was collected from the time of consent to 12-month post randomization.
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 11/87 | 5/33
Serious Adverse Events (participants affected / at risk) | 46/87 | 19/33
Other Adverse Events (participants affected / at risk) | 0/87 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=87) | Control Group (N=33)
Acute Coronary Syndromes (Cardiac disorders) | 2 (2) | 2 (2)
Arrhythmia - Atrial Fibrillation (Cardiac disorders) | 4 (4) | 1 (1)
Arrhythmia - Ventricular Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia - Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Spasm (Cardiac disorders) | 1 (1) | 0 (0)
ICD Device Shock (Cardiac disorders) | 1 (1) | 0 (0)
Heart Failure Exacerbation (Cardiac disorders) | 24 (24) | 11 (11)
Endocarditis (Cardiac disorders) | 0 (0) | 2 (2)
Sick Sinus Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Worsening of Mitral Regurgitation (Cardiac disorders) | 2 (2) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 4 (4) | 1 (1)
Infection (Infections and infestations) | 4 (4) | 2 (2)
Intracerebral Bleeding (Vascular disorders) | 0 (0) | 1 (1)
Lacunar Stroke (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2015-11-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT02325830/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT02325830/SAP_001.pdf